CLINICAL TRIAL: NCT05008900
Title: A Phase II Randomized Feasibility Study Comparing Early Salvage Radiotherapy Versus Surveillance With Delayed Repeat PSMA PET/CT Imaging in Patients Presenting With Early Biochemical Relapse of Prostate Cancer Following Radical Prostatectomy
Brief Title: Timing of Post-prostatectomy PSMA Imaging
Acronym: TOPP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-5040
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surveillance (Experimental): Patients with early biochemical relapse of prostate cancer following radical prostatectomy who have a PSA greater than or equal to 0.1 to less than 0.3 ng/mL with negative PSMA PET/CT will go on surveillance. Routine PSA will be conducted and a repeat PSMA PET/CT imaging will be conducted when the PSA rises to greater than 0.5 to less than 1.0 ng/mL.
  Interventions: Radiation: Salvage radiotherapy
- Salvage radiotherapy (No Intervention): Patients with early biochemical relapse of prostate cancer following radical prostatectomy who have a PSA of greater than or equal to 0.1 to less than 0.3 ng/mL with negative PSMA PET/CT will receive salvage radiotherapy to the prostate bed. This radiotherapy may or may not include the pelvic lymph nodes.

INTERVENTIONS:
Radiation: Salvage radiotherapy — Standard of care salvage radiotherapy to the prostate bed which may include the lymph nodes.
  Arms: Surveillance

SUMMARY:
The investigators will randomize patients presenting with early BCR with a negative baseline PSMA PET/CT, to upfront SRT or surveillance. Early BCR is defined as a PSA relapse of >0.1 to <0.3 ng/mL. Patients in the surveillance arm will be monitored with PSA every 3 months. A repeat PSMA PET/CT will be undertaken when the PSA reaches a target level of >0.5 to <1.0 ng/mL. Both early radiation treatment and surveillance with repeat PSMA PET/CT imaging are within patterns of practice locally; therefore, the investigators believe that there is clinical equipoise on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven prostate cancer
* pT1-T4 pN0/Nx cM0
* PSA at BCR >0.1 - <0.3 ng/mL post-radical prostatectomy
* PSMA PET/CT negative at BCR post radical prostatectomy
* Planned SRT to prostate bed +/- pelvic lymph nodes
* ECOG 0 or 1
* Age ≥ 18 years
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

Exclusion Criteria:

* Active or post prostatectomy androgen deprivation use
* Previous pelvic radiotherapy
* Other contraindications to radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Surveillance with delayed PSMA PET scan | 7 years
  This study will assess the feasibility of surveillance with delayed repeat PSMA PET/CT in patients with BCR of prostate cancer following radical prostatectomy with negative baseline PSMA PET/CT. A treating physician questionnaire will be completed prior to screening and enrollment, as well as PSA results every three months for surveillance patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada